CLINICAL TRIAL: NCT06201546
Title: Comparison of Abdominal Plane Blocks in Terms of Efficiency and Complications in Postoperative Pain Control in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Comparison of Abdominal Plane Blocks in Postoperative Pain Control in Patients Undergoing LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gamze Nur Teke, MD, assistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: gamzenurteke-1
Record Dates: First submitted 2023-02-25; First posted 2024-01-11 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgical Procedures; Anesthesia and Analgesia; Anesthesia, Regional
Keywords: LSG; TAP; m-TAPA; pain manangement; plane block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Clinical trial in which two groups of participants who are applied two type plane blocks. Group A; TAP block and group B; m-TAPA block. Effectiveness of blocks will be followed by appliying Pain Controlled Analgesia(PCA) and with pain scales as Visual Analog Scale(VAS) and Numerating Rate Scale.
Who Masked: Participant, Investigator
Masking Description: Due to the double-blind nature of the study, the outcome of the effectiveness of plane blocks will not be known by the anesthesiologist and the patient until the end of the study. Only the effectiveness of blocks will be followed by an another researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): Transversus Abdominal Plane Block aplied after LSG. In TAP block local anesthetic(%0,25 bupivacaine-20ml)will be administrated the between the transversus abdominis muscle and the internal abdominal muscle fascia.
  Interventions: Procedure: TAP block group
- m-TAPA block (Active Comparator): Modified-Thoracoabdominal Plane Block-pericondrial approach aplied after LSG. In m-TAPA block local anesthetic (0.25% bupivacaine-20ml) will be administrated between the transversus abdominis muscle and the internal abdominal muscle fascia under the costochondrial region.
  Interventions: Procedure: m-TAPA block group

INTERVENTIONS:
Procedure: TAP block group — TAP block will be administrated after LSG. In TAP block local anesthetic(%0,25 bupivacaine-20ml)will be administrated the between the transversus abdominis muscle and the internal abdominal muscle fascia.
  Arms: TAP block
Procedure: m-TAPA block group — m-TAPA block will be administrated after LSG. In m-TAPA block local anesthetic (0.25% bupivacaine-20ml) will be administrated between the transversus abdominis muscle and the internal abdominal muscle fascia under the costochondrial region
  Arms: m-TAPA block

SUMMARY:
The goal of this prospective observational study is compare in terms of efficiency and complications transversus abdominis plane (TAP) and Modified thoracoabdominal plane block-perichondrial approach (M-TAPA) blocks in patients undergoing laparoscopic sleeve gastrectomy. The investigators aims to examine whether M-TAPA block provides more effective analgesia than TAP block in upper abdomen surgeries, and whether there is any difference in terms of nausea- vomiting and need for additional analgesics. The participitans will be observed for postoperative 24 hours with numeric rating score (NRS), postoperative nausea-vomiting score (PNVS) and in terms of need for additional analgesic dose.

DETAILED DESCRIPTION:
After laparoscopic sleeve gastrectomy, patients have pain due to surgery. Different analgesic methods are preferred for pain relief. One of the methods used for this purpose is regional anesthesia. Modified thoracoabdominal plane block-perichondrial approach (M-TAPA) and transversus abdominis plane (TAP) block are also plan blocks used for this purpose. TAP block is formed by injecting local anesthetic into the neurofacial space between the transversus abdominis muscle and the internal oblique muscle through the Petit triangle in the lumbar region. TAP block creates dermatomal sensory block in the lower, lower thoracic and upper lumbar abdominal afferents. It is thought that the modified thoracoabdominal plane block-perichondrial approach (M-TAPA), which is a block frequently used in upper abdomen surgeries in recent years, can provide effective analgesia in LSG surgeries. M-TAPA block is created by administering local anesthetic between the transverse abdominis muscle and the internal oblique muscle with a single injection under the costal cartilage under ultrasound guidance. With M-TAPA, analgesia can be provided in thoracic 4 and thoracic 11-12 dermatomes.

Blocking of T4-12 nerve endings may be required in LSG surgeries, since gastric innervation and thoracic inlets are located in the upper abdomen dermatomes. In studies, the use of M-TAPA block in upper abdominal surgeries may be effective in the management of analgesia in participants. In this study the investigators aimed that, compression in terms of efficiency and complications TAP and M-TAPA blocks, who is undergoing laparoscopic sleeve gastrectomy. The investigators aims to examine whether M-TAPA block provides more effective analjesia than TAP block in upper abdomen surgeries, and whether there is any difference in terms of nausea- vomiting and need for additional analgesics. After obtaining ethical committee approval (12.01.2023/1), between January 26, 2023, and May 15, 2024, 60 patients undergoing laparoscopic sleeve gastrectomy with American Society of Anesthesiologists (ASA) II-III status provide informed consent. Participants who are planing to receive M-TAPA block defines as Group M-TAPA, and those who receive TAP block defines as Group TAP, with 30 patients in each group.The participitans will be observed for postoperative 24 hours with numeric rating score (NRS), postoperative nausea-vomiting score (PNVS) and in terms of need for additional analgesic dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65, including the ASA I-III group, who underwent laparoscopic sleeve gastrectomy by the General Surgery clinic between January 26, 2023 and May 15, 2023

Exclusion Criteria:

* Patients with coronary artery disease
* Patients with cerebrovascular disease
* Patients with peripheral artery disease
* History of chronic analgesic use
* Patients with coagulopathy
* Patients not between the ages of 18-65
* Patients with hepatic and/or renal insufficiency
* Patients with missing information in the information form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rate Score (NRS) | It will be evaluated with (which ), at PACU 5,15, 30th minutes and postoperative 1, 3, 6, 12, 24th hours
  NRS is a 0 to 10 scale that describes pain from good to worst.
Visual Analog Scale (VAS) | PACU 5,15, 30th minutes and postoperative 1, 3, 6, 12, 24th hours
  VAS is a 10-centimeter scale and is used to evaluate pain.
Pain Controlled Analgesia (PCA) | PACU 5,15, 30th minutes and postoperative 1, 3, 6, 12, 24th hours
  PCA is includes 300mg Tramadol/100 ml SF- no infusion, 5cc bolus, 15 minutes lock

SECONDARY OUTCOMES:
postoperative nausea and vomiting scale (PNV) | It will be evaluated with nause and vomiting score at PACU 5,15, 30th minutes and postoperative 1, 3, 6, 12, 24th hours
  PNV is a 0 to 4 scale that describes nausea and vomiting from good to worst.

CONTACTS AND LOCATIONS:
Overall Officials: arzu yıldırım ar, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Gamze Nur Teke, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838